CLINICAL TRIAL: NCT02722018
Title: A Phase I, Randomized, Open-Label, Single Center Study to Investigate the Effect of Formulation and Food on the Pharmacokinetics of GDC-0810 in Female Healthy Subjects on Non-Childbearing Potential
Brief Title: Study to Investigate the Effect of Formulation and Food on the Pharmacokinetics of GDC-0810
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GP29826; 2015-003730-27 (EudraCT Number)
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Healthy Volunteer

ARMS (3):
- Part 1: GDC-0810 dose level A - Low Fat Meal (Experimental): Participants will receive a single dose of GDC-0810 dose level A on Day 1 of each treatment period. GDC-0810 will be administered with low fat meal in the form of Phase II tablet or one of three Phase III prototype tablets (Prototype 1, 2 or 3) in a crossover fashion.
  Interventions: Drug: GDC-0810 Phase II Tablet; Drug: GDC-0810 Phase III Prototype Tablet
- Part 2 (Optional): GDC-0810 dose level A - Low Fat Meal (Experimental): Participants will receive a single dose of GDC-0810 dose level A on Day 1 of each treatment period. GDC-0810 will be administered with low fat meal in the form of Phase II tablet or one of two Phase III prototype tablets (Prototype 4 or 5) in a crossover fashion.
  Interventions: Drug: GDC-0810 Phase II Tablet; Drug: GDC-0810 Phase III Prototype Tablet
- Part 3: GDC-0810 dose level B - Low Fat Meal/Fasted (Experimental): Participants will receive a single dose of GDC-0810 dose level B on Day 1 of each treatment period. GDC-0810 will be administered with low fat meal or under fasted condition either as Phase II tablet (with low fat meal) or as the Phase III prototype tablet selected from Parts 1 or 2 (with low fat meal or under fasted conditions), in a crossover fashion.
  Interventions: Drug: GDC-0810 Phase II Tablet; Drug: GDC-0810 Phase III Prototype Tablet

INTERVENTIONS:
Drug: GDC-0810 Phase II Tablet — Participants will receive dose level A (in Parts 1 and 2) or dose level B (in Part 3) tablets.
Drug: GDC-0810 Phase III Prototype Tablet — Participants will receive dose level A (in Parts 1 and 2) or dose level B (in Part 3) tablets.

SUMMARY:
This is a phase 1, randomized, open-label, single center, crossover study to investigate the effect of formulation and food on the pharmacokinetics of GDC-0810 in female healthy participants of non-childbearing potential. This study is divided into three parts. Participants in each part will be randomized to one of three treatment sequences. Part 1 study in 4 periods will investigate the effect of formulation on the pharmacokinetics (PK) of GDC-0810 administered with low-fat food. Each participant in this part will receive a single dose of GDC-0810 dose level A following consumption of a low fat meal (30 minutes after the start of the meal) in each treatment period. Part 2 is an optional Phase I study in 3 periods to investigate the effect of formulation on the PK of GDC-0810 administered with low-fat food in healthy female participants of non-childbearing potential. Part 3 study in three periods will compare the PK of a Phase III prototype tablet formulation selected from Parts 1 and 2 of the study with the Phase II tablet formulation (both administered 30 minutes after the start of a low fat meal) at dose level B and to investigate the PK of the Phase III prototype formulation administered in the fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of non-childbearing potential including non-pregnant, non-lactating, and either postmenopausal or surgically sterile for at least 45 days post procedure
* Body mass index (BMI) range 18.0 to 32.0 kilograms per square meter (kg/m^2), inclusive
* In good health, as determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs, and clinical laboratory evaluations
* Receive an explanation of the mandatory pharmacogenomics (PgX) component of the study

Exclusion Criteria:

* Any history of endometrial polyps, endometrial cancer, atypical endometrial hyperplasia, or other endometrial disorders unless subjects have undergone total hysterectomy and there is no evidence of active disease
* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of any thrombophilic condition, inflammatory bowel disease, active bowel inflammation, chronic diarrhea, short bowel syndrome, and upper gastro-intestinal (GI) surgery including gastric resection
* Any history of venous thrombosis (including pulmonary embolism [PE])
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 90 days prior to Check-in (Day -1) in Period 1
* Use of systemic hormone replacement therapy within 1 year prior to Check-in (Day -1)
* History of use of tamoxifen, aromatase inhibitors, or any other endocrine agent for the treatment of breast cancer

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-09-13 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of GDC-0810 | Pre-dose (1 hour before dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16 hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3) of each treatment period
Time to Reach Cmax (Tmax) of GDC-0810 | Pre-dose (1 hour before dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16 hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3) of each treatment period
Area Under the Plasma Concentration Versus Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC0-t) of GDC-0810 | Pre-dose (1 hour before dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16 hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3) of each treatment period
Area Under the Plasma Concentration Versus Time Curve From Time Zero to Extrapolated Infinite Time (AUC0-inf) of GDC-0810 | Pre-dose (1 hour before dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16 hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3) of each treatment period
Apparent Terminal Elimination Rate Constant (lambda Z) of GDC-0810 | Pre-dose (1 hour before dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16 hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3) of each treatment period
Apparent Terminal Elimination Half-Life (t1/2) of GDC-0810 | Pre-dose (1 hour before dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16 hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3) of each treatment period
Apparent Oral Clearance (CL/F) of GDC-0810 | Pre-dose (1 hour before dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16 hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3) of each treatment period
Apparent Volume of Distribution (Vz/F) of GDC-0810 | Pre-dose (1 hour before dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16 hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3) of each treatment period
Relative Bioavailability Based on Cmax (Frel Cmax) of GDC-0810 (Test vs Reference) | Pre-dose (1 hour before dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16 hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3) of each treatment period
Relative Bioavailability Based on AUC0-t (Frel AUC0-t) of GDC-0810 (Test vs Reference) | Pre-dose (1 hour before dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16 hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3) of each treatment period
Relative Bioavailability Based on Cmax (Frel Cmax) of GDC-0810 (Fed vs Fasted) | Pre-dose (1 hour before dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16 hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3) of each treatment period
Relative Bioavailability Based on AUC0-t (Frel AUC0-t) of GDC-0810 (Fed vs Fasted) | Pre-dose (1 hour before dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16 hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3) of each treatment period

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Baseline up to 28 days after last GDC-0810 dose (Up to 57 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Quotient Clinical Ltd, Clinical Research Unit, Nottingham, United Kingdom